CLINICAL TRIAL: NCT05613972
Title: Using Integrated Suicide and Trauma Therapy to Reduce Suicide Risk Among Adults With a History of Childhood Trauma
Brief Title: Integrated Suicide & Trauma Therapy for Suicide Risk
Acronym: ISTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTT-01
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Trauma; Major Depressive Disorder
Keywords: Childhood trauma; Early life adversity; Adverse childhood experiences; Suicide intervention; Psychotherapy
MeSH Terms: conditions — Suicide; Wounds and Injuries; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Suicide and Trauma Therapy (BSTT) (Experimental): This novel suicide intervention integrates Brief Skills for Safer Learning (B-SfSL) with trauma therapy. ISTT incorporates the guiding principles of taking a non-pathologizing approach to treatment, emphasizing safety, attending to the therapeutic relationship, empowering clients, and incorporating solution-focused concepts.
  Interventions: Other: Integrated Suicide and Trauma Therapy

INTERVENTIONS:
Other: Integrated Suicide and Trauma Therapy — 12-week trauma therapy for suicide risk

SUMMARY:
The investigators have developed a novel suicide intervention, Integrated Suicide and Trauma Therapy (ISTT). ISTT combines Brief-Skills for Safer Living (Brief-SfSL)-a promising method to enhance coping skills and reduce suicidality-with a trauma therapy component to alleviate the specific impacts of childhood trauma on suicide risk. The aim of this pilot is to test 12-weeks of ISTT to alleviate suicide risk among individuals with a history of childhood trauma and current suicidality.

DETAILED DESCRIPTION:
In the last 10 years, despite available treatments, suicide rates have not significantly decreased, and individuals who have experienced any type of childhood maltreatment are at increased odds for suicide attempt. Effective suicide prevention requires learning skills to cope with suicidality in addition to addressing the antecedent factors that contribute to suicide risk. In the context of those with childhood trauma and suicidality, addressing antecedent factors may require treatments that target symptoms associated with developmental trauma. Thus, the investigators have developed an integrated suicide intervention, Integrated Suicide and Trauma Therapy (ISTT). ISTT combines Brief-Skills for Safer Living (Brief-SfSL)-a promising method to enhance coping skills and reduce suicidality-with a trauma therapy component to alleviate the specific impacts of childhood trauma on suicide risk. The aim of this pilot is to test 12-weeks of BSTT to alleviate suicide risk among individuals with a history of childhood trauma and current suicidality.

ELIGIBILITY:
Inclusion Criteria:

* Beck Scale for Suicidal Ideation > 10
* Presence of childhood trauma defined by a minimum moderate score on any of the Childhood Trauma Questionnaire subscales (emotional abuse, physical, abuse, sexual abuse, emotional neglect, and physical neglect
* Presence of any psychiatric diagnosis
* Ability to provide informed consent
* Not receiving other psychotherapy concurrently
* Ability to undergo psychotherapy in English

Exclusion Criteria:

* The presence of cognitive impairment that would limit consent or understanding of ISTT
* The presence of active psychosis
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicide Ideation (BSS) score | From baseline to 1 week post-therapy
  Beck Scale for Suicide Ideation is a 21-item self-report scale that quantifies suicidal ideation. Items are scored 0 to 2 and yield a total score ranging from 0 to 38. Higher scores reflect greater severity of suicidal ideation.
Feasibility and acceptability of ISTT | From baseline to 1 week post-therapy
  Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), Feasibility of Intervention Measure (FIM), in addition to a feedback survey and interview created in-house with questions designed to collect quantitative and qualitative feedback from participants with respect to the feasibility and acceptability of the BSTT intervention.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7-item scale (GAD-7) score | From baseline to 1-week post therapy
  The GAD-7 is a brief 7-item self-report scale measuring anxiety symptoms. Total scores range from 0 to 21, with higher scores reflecting more severe anxiety.
Change in Quick Inventory of Depressive Symptoms 16-item scale (QIDS) score | From baseline to 1 week post-therapy
  The QIDS is a 16-item validated depression scale. Total scores range from 0-27, with higher scores reflecting more severe depression.
Change in Difficulties in Emotion Regulation Scale 36-item scale (DERS) score | From baseline to 1 week post-therapy
  The DERS is a 36-item validated scale measuring six aspects of emotion regulation. The DERS is comprised of 6 subscales, where higher scores are reflective of greater difficulties in emotion regulation. The DERS is often analyzed by percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD,MACP,RP, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alloy LB, Abramson LY, Smith JM, Gibb BE, Neeren AM. Role of parenting and maltreatment histories in unipolar and bipolar mood disorders: mediation by cognitive vulnerability to depression. Clin Child Fam Psychol Rev. 2006 Mar;9(1):23-64. doi: 10.1007/s10567-006-0002-4. PMID 16718583
- [Background] Angelakis I, Gillespie EL, Panagioti M. Childhood maltreatment and adult suicidality: a comprehensive systematic review with meta-analysis. Psychol Med. 2019 May;49(7):1057-1078. doi: 10.1017/S0033291718003823. Epub 2019 Jan 4. PMID 30608046
- [Background] Bergmans Y, Links PS. Reducing potential risk factors for suicide-related behavior with a group intervention for clients with recurrent suicide-related behavior. Ann Clin Psychiatry. 2009 Jan-Mar;21(1):17-25. PMID 19239829
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Berube A, Turgeon J, Blais C, Fiset D. Emotion Recognition in Adults With a History of Childhood Maltreatment: A Systematic Review. Trauma Violence Abuse. 2023 Jan;24(1):278-294. doi: 10.1177/15248380211029403. Epub 2021 Jul 9. PMID 34238064
- [Background] Bremness A, Polzin W. Commentary: Developmental Trauma Disorder: A Missed Opportunity in DSM V. J Can Acad Child Adolesc Psychiatry. 2014 May;23(2):142-5. No abstract available. PMID 24872830
- [Background] Briggs S, Netuveli G, Gould N, Gkaravella A, Gluckman NS, Kangogyere P, Farr R, Goldblatt MJ, Lindner R. The effectiveness of psychoanalytic/psychodynamic psychotherapy for reducing suicide attempts and self-harm: systematic review and meta-analysis. Br J Psychiatry. 2019 Jun;214(6):320-328. doi: 10.1192/bjp.2019.33. Epub 2019 Feb 28. PMID 30816079
- [Background] Brom D, Stokar Y, Lawi C, Nuriel-Porat V, Ziv Y, Lerner K, Ross G. Somatic Experiencing for Posttraumatic Stress Disorder: A Randomized Controlled Outcome Study. J Trauma Stress. 2017 Jun;30(3):304-312. doi: 10.1002/jts.22189. Epub 2017 Jun 6. PMID 28585761
- [Background] Bryan CJ, Clemans TA, Hernandez AM, Mintz J, Peterson AL, Yarvis JS, Resick PA; STRONG STAR Consortium. EVALUATING POTENTIAL IATROGENIC SUICIDE RISK IN TRAUMA-FOCUSED GROUP COGNITIVE BEHAVIORAL THERAPY FOR THE TREATMENT OF PTSD IN ACTIVE DUTY MILITARY PERSONNEL. Depress Anxiety. 2016 Jun;33(6):549-57. doi: 10.1002/da.22456. Epub 2015 Dec 4. PMID 26636426
- [Background] Cao H, Ma R, Li X, Liang Y, Wu Q, Chi P, Li JB, Zhou N. Childhood Emotional Maltreatment and Adulthood Romantic Relationship Well-Being: A Multilevel, Meta-Analytic Review. Trauma Violence Abuse. 2022 Jul;23(3):778-794. doi: 10.1177/1524838020975895. Epub 2020 Dec 3. PMID 33267741
- [Background] Cloitre M, Courtois CA, Charuvastra A, Carapezza R, Stolbach BC, Green BL. Treatment of complex PTSD: results of the ISTSS expert clinician survey on best practices. J Trauma Stress. 2011 Dec;24(6):615-27. doi: 10.1002/jts.20697. Epub 2011 Dec 6. PMID 22147449
- [Background] Copeland WE, Shanahan L, Hinesley J, Chan RF, Aberg KA, Fairbank JA, van den Oord EJCG, Costello EJ. Association of Childhood Trauma Exposure With Adult Psychiatric Disorders and Functional Outcomes. JAMA Netw Open. 2018 Nov 2;1(7):e184493. doi: 10.1001/jamanetworkopen.2018.4493. PMID 30646356
- [Background] Coventry PA, Meader N, Melton H, Temple M, Dale H, Wright K, Cloitre M, Karatzias T, Bisson J, Roberts NP, Brown JVE, Barbui C, Churchill R, Lovell K, McMillan D, Gilbody S. Psychological and pharmacological interventions for posttraumatic stress disorder and comorbid mental health problems following complex traumatic events: Systematic review and component network meta-analysis. PLoS Med. 2020 Aug 19;17(8):e1003262. doi: 10.1371/journal.pmed.1003262. eCollection 2020 Aug. PMID 32813696
- [Background] Cruz D, Lichten M, Berg K, George P. Developmental trauma: Conceptual framework, associated risks and comorbidities, and evaluation and treatment. Front Psychiatry. 2022 Jul 22;13:800687. doi: 10.3389/fpsyt.2022.800687. eCollection 2022. PMID 35935425
- [Background] Doyle C, Cicchetti D. From the Cradle to the Grave: The Effect of Adverse Caregiving Environments on Attachment and Relationships Throughout the Lifespan. Clin Psychol (New York). 2017 Jun;24(2):203-217. doi: 10.1111/cpsp.12192. Epub 2017 Apr 11. PMID 28924334
- [Background] Fereidouni Z, Behnammoghadam M, Jahanfar A, Dehghan A. The Effect of Eye Movement Desensitization and Reprocessing (EMDR) on the severity of suicidal thoughts in patients with major depressive disorder: a randomized controlled trial. Neuropsychiatr Dis Treat. 2019 Aug 27;15:2459-2466. doi: 10.2147/NDT.S210757. eCollection 2019. PMID 31695382
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Fischer A, Rosner R, Renneberg B, Steil R. Suicidal ideation, self-injury, aggressive behavior and substance use during intensive trauma-focused treatment with exposure-based components in adolescent and young adult PTSD patients. Borderline Personal Disord Emot Dysregul. 2022 Jan 3;9(1):1. doi: 10.1186/s40479-021-00172-8. PMID 34974844
- [Background] Freeman A, Mergl R, Kohls E, Szekely A, Gusmao R, Arensman E, Koburger N, Hegerl U, Rummel-Kluge C. A cross-national study on gender differences in suicide intent. BMC Psychiatry. 2017 Jun 29;17(1):234. doi: 10.1186/s12888-017-1398-8. PMID 28662694
- [Background] Grummitt LR, Kreski NT, Kim SG, Platt J, Keyes KM, McLaughlin KA. Association of Childhood Adversity With Morbidity and Mortality in US Adults: A Systematic Review. JAMA Pediatr. 2021 Dec 1;175(12):1269-1278. doi: 10.1001/jamapediatrics.2021.2320. PMID 34605870
- [Background] Guo Y, Ji Y, Huang Y, Jin M, Lin Y, Chen Y, Zhang L, Zhu C, Yu F, Wang K. The Relationship Between Suicidal Ideation and Parental Attachment Among Adolescents: The Mediator of Anhedonia and Peer Attachment. Front Psychol. 2021 Oct 18;12:727088. doi: 10.3389/fpsyg.2021.727088. eCollection 2021. PMID 34733205
- [Background] Hakamata Y, Suzuki Y, Kobashikawa H, Hori H. Neurobiology of early life adversity: A systematic review of meta-analyses towards an integrative account of its neurobiological trajectories to mental disorders. Front Neuroendocrinol. 2022 Apr;65:100994. doi: 10.1016/j.yfrne.2022.100994. Epub 2022 Mar 21. PMID 35331780
- [Background] Harned MS, Korslund KE, Linehan MM. A pilot randomized controlled trial of Dialectical Behavior Therapy with and without the Dialectical Behavior Therapy Prolonged Exposure protocol for suicidal and self-injuring women with borderline personality disorder and PTSD. Behav Res Ther. 2014 Apr;55:7-17. doi: 10.1016/j.brat.2014.01.008. Epub 2014 Feb 11. PMID 24562087
- [Background] Hawton K, Casanas I Comabella C, Haw C, Saunders K. Risk factors for suicide in individuals with depression: a systematic review. J Affect Disord. 2013 May;147(1-3):17-28. doi: 10.1016/j.jad.2013.01.004. Epub 2013 Feb 12. PMID 23411024
- [Background] Herzog JI, Schmahl C. Adverse Childhood Experiences and the Consequences on Neurobiological, Psychosocial, and Somatic Conditions Across the Lifespan. Front Psychiatry. 2018 Sep 4;9:420. doi: 10.3389/fpsyt.2018.00420. eCollection 2018. PMID 30233435
- [Background] Itzhaky L, Gratch I, Galfalvy H, Keilp JG, Burke AK, Oquendo MA, Mann JJ, Stanley BH. Psychosocial risk factors and outcomes associated with suicide attempts in childhood: A retrospective study. J Psychiatr Res. 2020 Jun;125:129-135. doi: 10.1016/j.jpsychires.2020.03.008. Epub 2020 Mar 18. PMID 32278224
- [Background] Karatzias T, Murphy P, Cloitre M, Bisson J, Roberts N, Shevlin M, Hyland P, Maercker A, Ben-Ezra M, Coventry P, Mason-Roberts S, Bradley A, Hutton P. Psychological interventions for ICD-11 complex PTSD symptoms: systematic review and meta-analysis. Psychol Med. 2019 Aug;49(11):1761-1775. doi: 10.1017/S0033291719000436. Epub 2019 Mar 12. PMID 30857567
- [Background] Michel K, Valach L, Gysin-Maillart A. A Novel Therapy for People Who Attempt Suicide and Why We Need New Models of Suicide. Int J Environ Res Public Health. 2017 Mar 1;14(3):243. doi: 10.3390/ijerph14030243. PMID 28257071
- [Background] Miniati M, Callari A, Pini S. Adult Attachment Style and Suicidality. Psychiatr Danub. 2017 Sep;29(3):250-259. doi: 10.24869/psyd.2017.250. PMID 28949306
- [Background] Mitchell TO, Li L. State-Level Data on Suicide Mortality During COVID-19 Quarantine: Early Evidence of a Disproportionate Impact on Racial Minorities. Psychiatry Res. 2021 Jan;295:113629. doi: 10.1016/j.psychres.2020.113629. Epub 2020 Dec 3. PMID 33290944
- [Background] Miu AC, Szentagotai-Tatar A, Balazsi R, Nechita D, Bunea I, Pollak SD. Emotion regulation as mediator between childhood adversity and psychopathology: A meta-analysis. Clin Psychol Rev. 2022 Apr;93:102141. doi: 10.1016/j.cpr.2022.102141. Epub 2022 Feb 21. PMID 35219929
- [Background] Novick AM, Levandowski ML, Laumann LE, Philip NS, Price LH, Tyrka AR. The effects of early life stress on reward processing. J Psychiatr Res. 2018 Jun;101:80-103. doi: 10.1016/j.jpsychires.2018.02.002. Epub 2018 Feb 13. PMID 29567510
- [Background] O'Connor RC, Kirtley OJ. The integrated motivational-volitional model of suicidal behaviour. Philos Trans R Soc Lond B Biol Sci. 2018 Sep 5;373(1754):20170268. doi: 10.1098/rstb.2017.0268. PMID 30012735
- [Background] Oon-Arom A, Wongpakaran T, Satthapisit S, Saisavoey N, Kuntawong P, Wongpakaran N. Suicidality in the elderly: Role of adult attachment. Asian J Psychiatr. 2019 Aug;44:8-12. doi: 10.1016/j.ajp.2019.07.014. Epub 2019 Jul 5. PMID 31302442
- [Background] Oral R, Ramirez M, Coohey C, Nakada S, Walz A, Kuntz A, Benoit J, Peek-Asa C. Adverse childhood experiences and trauma informed care: the future of health care. Pediatr Res. 2016 Jan;79(1-2):227-33. doi: 10.1038/pr.2015.197. Epub 2015 Oct 13. PMID 26460523
- [Background] Pirkis J, John A, Shin S, DelPozo-Banos M, Arya V, Analuisa-Aguilar P, Appleby L, Arensman E, Bantjes J, Baran A, Bertolote JM, Borges G, Brecic P, Caine E, Castelpietra G, Chang SS, Colchester D, Crompton D, Curkovic M, Deisenhammer EA, Du C, Dwyer J, Erlangsen A, Faust JS, Fortune S, Garrett A, George D, Gerstner R, Gilissen R, Gould M, Hawton K, Kanter J, Kapur N, Khan M, Kirtley OJ, Knipe D, Kolves K, Leske S, Marahatta K, Mittendorfer-Rutz E, Neznanov N, Niederkrotenthaler T, Nielsen E, Nordentoft M, Oberlerchner H, O'Connor RC, Pearson M, Phillips MR, Platt S, Plener PL, Psota G, Qin P, Radeloff D, Rados C, Reif A, Reif-Leonhard C, Rozanov V, Schlang C, Schneider B, Semenova N, Sinyor M, Townsend E, Ueda M, Vijayakumar L, Webb RT, Weerasinghe M, Zalsman G, Gunnell D, Spittal MJ. Suicide trends in the early months of the COVID-19 pandemic: an interrupted time-series analysis of preliminary data from 21 countries. Lancet Psychiatry. 2021 Jul;8(7):579-588. doi: 10.1016/S2215-0366(21)00091-2. Epub 2021 Apr 13. PMID 33862016
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Roy A. Relationship of childhood trauma to age of first suicide attempt and number of attempts in substance dependent patients. Acta Psychiatr Scand. 2004 Feb;109(2):121-5. doi: 10.1046/j.0001-690x.2003.00234.x. PMID 14725593
- [Background] Rozek DC, Baker SN, Rugo KF, Steigerwald VL, Sippel LM, Holliday R, Roberge EM, Held P, Mota N, Smith NB. Addressing co-occurring suicidal thoughts and behaviors and posttraumatic stress disorder in evidence-based psychotherapies for adults: A systematic review. J Trauma Stress. 2022 Apr;35(2):729-745. doi: 10.1002/jts.22774. Epub 2021 Dec 31. PMID 34973046
- [Background] Schottenbauer MA, Glass CR, Arnkoff DB, Tendick V, Gray SH. Nonresponse and dropout rates in outcome studies on PTSD: review and methodological considerations. Psychiatry. 2008 Summer;71(2):134-68. doi: 10.1521/psyc.2008.71.2.134. PMID 18573035
- [Background] Smith KE, Pollak SD. Early life stress and development: potential mechanisms for adverse outcomes. J Neurodev Disord. 2020 Dec 16;12(1):34. doi: 10.1186/s11689-020-09337-y. PMID 33327939
- [Background] Stagaki M, Nolte T, Feigenbaum J, King-Casas B, Lohrenz T, Fonagy P; Personality and Mood Disorder Research Consortium; Montague PR. The mediating role of attachment and mentalising in the relationship between childhood maltreatment, self-harm and suicidality. Child Abuse Negl. 2022 Jun;128:105576. doi: 10.1016/j.chiabu.2022.105576. Epub 2022 Mar 18. PMID 35313127
- [Background] Turecki G, Brent DA. Suicide and suicidal behaviour. Lancet. 2016 Mar 19;387(10024):1227-39. doi: 10.1016/S0140-6736(15)00234-2. Epub 2015 Sep 15. PMID 26385066
- [Background] Ueda M, Nordstrom R, Matsubayashi T. Suicide and mental health during the COVID-19 pandemic in Japan. J Public Health (Oxf). 2022 Aug 25;44(3):541-548. doi: 10.1093/pubmed/fdab113. PMID 33855451
- [Background] Valle LA, Silovsky JF. Attributions and adjustment following child sexual and physical abuse. Child Maltreat. 2002 Feb;7(1):9-25. doi: 10.1177/1077559502007001002. PMID 11838520
- [Background] Ward-Ciesielski EF, Wilks CR. Conducting Research with Individuals at Risk for Suicide: Protocol for Assessment and Risk Management. Suicide Life Threat Behav. 2020 Apr;50(2):461-471. doi: 10.1111/sltb.12602. Epub 2019 Nov 8. PMID 31702077
- [Background] Zortea TC, Dickson A, Gray CM, O'Connor RC. Associations between experiences of disrupted attachments and suicidal thoughts and behaviours: An interpretative phenomenological analysis. Soc Sci Med. 2019 Aug;235:112408. doi: 10.1016/j.socscimed.2019.112408. Epub 2019 Jul 10. PMID 31323541
- [Background] Zortea TC, Gray CM, O'Connor RC. The Relationship Between Adult Attachment and Suicidal Thoughts and Behaviors: A Systematic Review. Arch Suicide Res. 2021 Jan-Mar;25(1):38-73. doi: 10.1080/13811118.2019.1661893. Epub 2019 Sep 23. PMID 31545148